CLINICAL TRIAL: NCT04462159
Title: Young Patients With Coronary Heart Disease Trial- Assessment of Risk Factors and the Impact of a Risk Reduction Program
Brief Title: The Young Heart Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-0073
Record Dates: First submitted 2020-02-20; First posted 2020-07-08 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Atherosclerotic Cardiovascular Disease; Coronary Artery Disease
Keywords: cardiovascular disease; coronary artery disease; myocardial infarction; risk factors; gender disparities; novel biomarkers; lifestyle behaviors
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Cardiovascular Diseases; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risk Reduction Program (Experimental): All participants will receive education about the process of atherosclerosis, risk factors contributing to the disease and specific risk factor goals for each patient for the 6 month program. The patients will then be part of a bimonthly 6 month cardiovascular risk reduction program that will offer both a nutritional program with teaching kitchen component, and exercise instruction lead by an exercise physiologist. Psychological support will be provided to address stress that impairs quality of life, depression or anxiety to fully optimize the lifestyle component.
  Interventions: Behavioral: Risk Reduction Program

INTERVENTIONS:
Behavioral: Risk Reduction Program — Education, exercise, teaching kitchen and nutrition, and psychological support

SUMMARY:
The purpose of our project is to better understand the characteristics of the young patients with coronary artery disease presenting for cardiac catheterization at our institution and to put forth a program to optimize their risk factors with a focus on gender differences. We will assess traditional and non-traditional risk factors, as well as genetics and environment. These characteristics will be compared by gender to determine unique factors related to women that could subsequently be targeted. The program will begin with universal education about the process of atherosclerosis, risk factors contributing to the disease and specific risk factor goals for each patient for the 6 month program. The patients will then be part of a bimonthly 6 month cardiovascular risk reduction program that will offer both a nutritional program with teaching kitchen component, and exercise instruction lead by an exercise physiologist. Psychological support will be provided to address stress that impairs quality of life, depression or anxiety to fully optimize the lifestyle component. These sessions will be done virtually in order to comply with social distancing until in person sessions can resume.

The investigational endpoints of this program will include a variety of cardiovascular disease (CVD) risk factors, biomarkers, lifestyle behaviors, quality of life and guideline-based medical regimen. At the end of this phase, we aim to both better understand differences in risk factors and the interventions with the biggest impact in terms of risk factor optimization in men vs. women.

DETAILED DESCRIPTION:
After enrollment, participants will meet with researchers where baseline character-istics will be obtained including biometrics such as weight, height, blood pressure, abdominal circumference, etc., as well as a questionnaire that will include validat-ed screening tools for the screening for depression, anxiety, and stress, which are considered non-traditional risk factors for heart disease. The questionnaire will also include other aspects of the participant's lifestyle that could help better understand their risk for heart disease. This questionnaire will be available to be filled out on paper, via email which will be linked with REDCap, and in a tablet provided by our team with the data also being uploaded directly to REDCap.

Blood will also be collected by venipuncture (approximately 12milliliters, 6-8mL for standard of care labs, and 3-4mL for research labs) to assess inflammatory markers, lipids and glucose levels. If based on this initial screening, participants are thought to be at high risk for genetic disease, which likely predisposed them to develop heart disease, they will be offered genetic testing as part of their routine clinical care outside of this research, and an additional consent form will then be provided. We are planning to only recommend genetic testing as per clinical care in those for whom it is recommended by clinical guidelines. When a patient is deemed eligible from a clinical standpoint, they will be referred to our cardio ge-nomics team and be consented as per their clinical protocols and samples, either saliva or blood acquired by venipuncture (about 5ml), will be obtained. Source of sample will be determined by cardio genomics team and this will also fall under their standard of care. If the patient is being enrolled in the outpatient setting and has lab work within the past month, assuming no changes have been made to lipid lowering therapies during that time, we will only need to draw 3-4mL for research labs and possibly one additional tube for Lipoprotein A, as it is not commonly in-cluded in basic lab work.

During their initial consultation while in the hospital, their individual risk would be assessed and the patient will receive counseling on how to further improve said risk. These goals will be reinforced and measures to ensure those goals are met will be implemented when the patient comes to clinic within 2 weeks from their cardiac catheterization. During that visit, they will also be educated on the process of heart disease. Frequency of follow up in clinic will be determined on an individual basis based on individual risk factors, however, all patients are expected to be seen for a minimum of 3 times during those 6 months.

Soon after seeing us for that initial visit in clinic, the group risk reduction program will begin and will last for 6 months with 2 sessions per month (every other week), out of which participants will be required to attend at least 6 for maximum benefit. The sessions will include an exercise and nutrition program.

The nutrition program will be given by a Registered Dietitian Nutritionist and it will consist of a 60min session that will include about 10-15min education, 30min for a cooking demonstration where participants will be able to participate in the process of making heart healthy foods, and 10-15min for questions and answers. Food al-lergies will be reviewed prior to initiation of each session.

The exercise portion of the program will be led by a RRCA Level 1 Certified Coach from Achilles International and the exercise will be low level exercise, at a level lower than even cardiac rehabilitation, which is usually recommended for patients after cardiac procedures. Regardless, the patient's cardiologist will indicate in writ-ing that it is safe to proceed with these sessions, which will be a 60min session provided by an exercise specialist.

Both nutrition and exercise sessions will occur between 5:30-6:30pm or 6pm-7pm at the Friedman Institute for Diabetes, and if the weather allows, some of the exer-cise sessions will be at Central Park. If needed, participants can also see a psy-chologist. Once the risk reduction program has ended, within a month we will re-evaluate the participants, repeat the initial questionnaire (excluding the demo-graphic data, past medical history and family history sections) and repeat blood work, with the exception of referral for genetic testing.

The registered dietitian and exercise coach are not considered investigators on this study as they will be performing their routine job function and will not be giving any new or different information to the participants of this study than what they would give to any other person joining them who are not part of this study. Addi-tionally, they will not be collecting any data either.

Results will be analyzed by gender with the intention to assess if some characteris-tics are unique to women compared to men, and the impact of the program on risk factors will also be assessed. Participants will also be called by one of the re-searchers about 1 month after the program has finished to assess if any changes in their lifestyle have persisted after the program, and once a year to follow up on cardiovascular events for 5yrs.

Addendum:

The Young Heart Study was designed to help subjects identify, educate, and reduce their risk of cardiovascular disease. The original structure of the study was to hold in-person sessions geared towards mental health, nutrition, and exercise. The widespread impact of COVID-19 forced the research team to pivot from the previ-ous model and include innovative virtual supplemental content.

The Young Heart Study has developed 3 instructional videos in the areas of mental health, nutrition, and exercise. These videos will be used in addition to physically distanced in-person events in accordance with CDC recommendations. The virtual content will not replace the original in-person events and is to be used in addition to the original study procedures.

The revised protocol is for ALL subjects to watch the video content and answer a short experiential survey (included on separate document). This survey will help the research team gauge impact of the videos and determine use case for the remain-der of the study.

The post-study survey provided after the 6 month period will be used to gauge perceived improvement by participant, improve relevant data collection, and add additional qualitative information to study team.

ELIGIBILITY:
Inclusion Criteria:

* Patient with atherosclerotic cardiovascular disease

Exclusion Criteria:

* Age 60 years or older
* Physical limitation that will prevent them from being part of the exercise part of the study
* Given that all the sessions will be given in English, participants not fluent in English will be excluded

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiovascular (CV) Risk Factor - Cholesterol levels | 6 months
  Will assess changes pre and post intervention in Low Density Lipoprotein Cholesterol level (measured in mg/dL)
Change in CV Risk Factor - Blood pressure | 6 months
  Will assess changes pre and post intervention in blood pressure (mmHg)
Change in CV Risk Factor - Glucometabolic state (A1C) | 6 months
  Will assess changes pre and post intervention in glycemic control measured by the hemoglobin A1C (%)
Change in CV Risk Factor - Smoking Status | 6 months
  Will assess changes pre and post intervention in smoking status (including quantity of cigarettes)
Change in CV Risk Factor - Physical activity/inactivity | 6 months
  Will assess changes pre and post intervention in physical activity which will be done through a questionnaire where participants will report the frequency and intensity of exercise
Change in CV Risk Factor - Overweight/Obesity | 6 months
  Will assess changes in weight by weighing patients on initial visit and again at follow-up. This value will be used in combination with patient's height to evaluate changes in body mass index.
Change in CV Risk Factors - Diet | 6 months
  Will assess changes pre and post intervention in diet which will be done via a food intake questionnaire
Change in CV Risk Factors - TMAO levels | 6 months
  Will assess changes pre and post intervention in trimethylamine N-oxide (TMAO) levels (microM)
Change in CV Risk Factors - hs-CRP levels | 6 months
  Will assess changes pre and post intervention in high sensitive C-reactive protein (hs-CRP) measured in mg/L
Change in Quality of Life Score | 6 months
  Surveys of Quality of Life and emotional well-being will be given at baseline and again at the end of the program

SECONDARY OUTCOMES:
Number of Cardiovascular events | 5 years
  Cardiovascular events assessed by a yearly phone call to the patient for up to 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Eugenia Gianos, MD, Principal Investigator — Northwell Health
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No